CLINICAL TRIAL: NCT02942693
Title: A Phase II Randomized Trial of Efficacy and Safety of Particle Therapy With or Without Apatinib as Induction Therapy for Treatment of Head and Neck Adenoid Cystic Carcinoma
Brief Title: Trail Evaluating Particle Therapy With or Without Apatinib for H&N Adenoid Cystic Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Jiade J. Lu, Executive Vice President of Shanghai Proton and Heavy Ion Center, Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HNCNS-2016-08
Record Dates: First submitted 2016-10-18; First posted 2016-10-24 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: Apatinib; Particle therapy
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apatinib with Particle Therapy (Experimental): Participants will receive apatinib (0.5g, daily) for 6 weekly followed by particle radiotherapy (proton: 56 GyE/28 Fx, plus carbon: 15 GyE/5 Fx for boost).
  Interventions: Drug: Apatinib; Radiation: Particle Therapy
- Particle Therapy (Experimental): Participants will receive particle radiotherapy alone (proton: 56 GyE/28 Fx, plus carbon: 15 GyE/5 Fx for boost).
  Interventions: Radiation: Particle Therapy

INTERVENTIONS:
Drug: Apatinib — Apatinib will be used as induction therapy in experimental arm.
  Arms: Apatinib with Particle Therapy
Radiation: Particle Therapy — Same total dose and fractionation will be used in both arms.

SUMMARY:
It is a randomized phase II study to determine the efficacy and safety of particle therapy with or without apatinib as induction therapy for the treatment of head and neck adenoid cystic carcinoma. Participants will be randomized to arm 1: receiving apatinib for 6 weekly followed by particle radiotherapy; arm 2: particle radiotherapy alone.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy and safety of particle therapy with or without apatinib as induction therapy for the treatment of head and neck adenoid cystic carcinoma. It is a randomized phase II clinical trial with single phase and 2 experimental arms. Participants will be randomized to arm 1, receiving apatinib (0.5g, daily) for 6 weekly followed by particle radiotherapy (proton: 56 GyE/28 Fx, plus carbon: 15 GyE/5 Fx for boost); arm 2: particle radiotherapy alone (proton: 56 GyE/28 Fx, plus carbon: 15 GyE/5 Fx for boost). The short term response will be evaluated using RECIST criteria. And the acute and late toxicities will be evaluated according to NCI CTCAE v4.03.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed ACC
* Inoperable disease or postoperative residual disease detected by imaging studies
* Age ≥ 18 and ≤ 65 years of age
* ECOG < 2, no significant active concurrent medical illnesses
* Adequate laboratory values within 30 dyas of enrollment to study defined as follows: N > 2000/mm^3; PLT > 100,000/mm^3; total bilirubin < 1.5mg/dl; AST/ALT < 1.5 ULN; SCr < 1.5mg/dl; CCR > 60ml/min
* Willing to accept adequate contraception for women with childbearing potential
* Ability to understand character and individual consequences of the clinical trial
* Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial

Exclusion Criteria:

* Presence of distant metastasis
* Pregnant or lactating women
* A diagnosis of malignancy other than CIS of the cervix, BCC and SCC of the skin within the past 5 years
* Refusal of the patient to participate into the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Short-term treatment response of all patients | Three months after completion of particle therapy.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI CTCAE v4.03 | Time interval from start to 3 months after completion of particle therapy.
Overall survival of all patients | From the diagnosis of H&N adenoid cystic carcinoma, a median of 3 years.
Progression-free survival of all patients | From the completion of the particle therapy, a median of 3 years.
Local progression-free survival of all patients | From the completion of the particle therapy, a median of 3 years.
Distant metastasis-free survival of all patients | From the completion of the particle therapy, a median of 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jiade J Lu, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center,Shanghai, SPHIC
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided